CLINICAL TRIAL: NCT05011955
Title: Brief Online Mindfulness and Intercare Based Intervention for Medicine Students (MIIM)
Brief Title: Mindfulness and Intercare Based Intervention for Medicine Students (MIIM)
Acronym: MIIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Diego Portales (Other)
Responsible Party: Principal Investigator, Francisco Javier Villalon Lopez, Principal Investigator, University Diego Portales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-2020
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Depressive Symptoms; Mental Health Wellness 1; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness, compassion and intercare based Intervention (Experimental): Four week, one hour peer week, online group intervention plus home work based on mindfulness, compassion and intercare based programs.
  Interventions: Behavioral: Mindfulness, compassion and intercare based Intervention; Other: General curricular intervention
- Psychoeducational based intervention (Active Comparator): Four week, one hour peer week, online group intervention plus home work based on psychoeducation about stress, anxiety, selfcare and effective communication.
  Interventions: Behavioral: Psychoeducational based intervention; Other: General curricular intervention
- General curricular intervention (Other): All participants were offered psychological sessions if a high score on depression or anxiety symptoms were detected. Participants also have academic breaks of two week per semester, apart from holidays, and academic flexibility in submitting work, attending practical activities and taking exams.
  Interventions: Other: General curricular intervention

INTERVENTIONS:
Behavioral: Mindfulness, compassion and intercare based Intervention — The mindfulness based intervention was a short version of the Mindfulness based intercare program (IBAP). The intervention consists of four synchronic group sessions via ZOOM of one hour each, one peer week and home practice. A total of four groups were conducted of 15 students each.
  The IBAP program was inspired by first and second generation mindfulness based interventions, such as Mindfulness based cognitive training, Self-Compassion and Cognitive based Compassion training. Also compassionate communication, conservation of resource theory and habits theory.
  Each module consists in meditation practices, inquiry and self or group reflections on different topics such as mindfulness, automatic pilot, mind wandering , acceptance, gratitude and compassion, care resources and intercare.
  Arms: Mindfulness, compassion and intercare based Intervention
Behavioral: Psychoeducational based intervention — Four week, one hour peer week, online group intervention plus home work base on psychoeducation about stress, anxiety, selfcare and effective communication. Plus general curricular intervention. Delivered by psychologist.
  Arms: Psychoeducational based intervention
Other: General curricular intervention — All participants were offered psychological sessions if a high score on depression or anxiety symptoms were detected. Psychological sessions consists of 4 to 8 sessions with specific objectives and then referral to continue the mental health process according to the student's welfare system.
  Participants also have academic breaks of two week per semester, apart from holidays, and academic flexibility in submitting work, attending practical activities and taking exams.

SUMMARY:
The effects of Coronavirus Disease (COVID-19) pandemic on health, economy and social network has an impact on mental health, specially students. The aim of the study was to evaluate the effectiveness of a brief online mindfulness, compassion and intercare based intervention in medicine students in Santiago de Chile.

Randomized controlled trial was conducted. Enrolled participants were randomly assigned to 1) a mindfulness, compassion and intercare based intervention, 2) a psychoeducational intervention or 3) waiting list. Both intervention lasted 1 hour per week for 4 weeks. Academic flexibility, breaks and individual psychological help was offered to the whole group. An online assessment of well being, anxiety and depression symptoms was completed at the beginning, 1 month and 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Medicine Students
* 1st to 7th class year

Exclusion Criteria:

* Recent Grief
* Severe acute depression disorder
* Active suicidal ideation
* Active Psychosis
* Active addiction
* Post Traumatic Stres Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, Female, Non Binary, Other
Enrollment: 360 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Depression symptoms - Patient Health Questionnaire - 9 (PHQ9) | Baseline
  Depression symptoms were evaluated using the Patient Health Questionnaire - 9 (PHQ9), which its used for depression screening with a sensibility and specificity of 88% y 92%. It contains 9 items on a 5-point Likert scale (0-4) to evaluate frequency of symptoms from "Never" to "Almost every day".
Depression symptoms - Patient Health Questionnaire - 9 (PHQ9) | 1 month - after intervention
  Depression symptoms were evaluated using the Patient Health Questionnaire - 9 (PHQ9), which its used for depression screening with a sensibility and specificity of 88% y 92%. It contains 9 items on a 5-point Likert scale (0-4) to evaluate frequency of symptoms from "Never" to "Almost every day".
Depression symptoms - Patient Health Questionnaire - 9 (PHQ9) | 3 month
  Depression symptoms were evaluated using the Patient Health Questionnaire - 9 (PHQ9), which its used for depression screening with a sensibility and specificity of 88% y 92%. It contains 9 items on a 5-point Likert scale (0-4) to evaluate frequency of symptoms from "Never" to "Almost every day".
Anxiety symptoms - General Anxiety Disorder 7 (GAD-7) | Baseline
  Anxiety symptoms were evaluated using the General Anxiety Disorder 7 (GAD-7) validated on Spanish population for anxiety disorder screening with a a sensibility and specificity of 86,8% and 93,4%. It contains 7 items on a 5-point Likert scale (0-3) to evaluate frequency of symptoms from "Never" to "Almost every day".
Anxiety symptoms - General Anxiety Disorder 7 (GAD-7) | 1 month - after intervention
  Anxiety symptoms were evaluated using the General Anxiety Disorder 7 (GAD-7) validated on Spanish population for anxiety disorder screening with a a sensibility and specificity of 86,8% and 93,4%. It contains 7 items on a 5-point Likert scale (0-3) to evaluate frequency of symptoms from "Never" to "Almost every day".
Anxiety symptoms - General Anxiety Disorder 7 (GAD-7) | 3 month
  Anxiety symptoms were evaluated using the General Anxiety Disorder 7 (GAD-7) validated on Spanish population for anxiety disorder screening with a a sensibility and specificity of 86,8% and 93,4%. It contains 7 items on a 5-point Likert scale (0-3) to evaluate frequency of symptoms from "Never" to "Almost every day".

SECONDARY OUTCOMES:
Mental Health - Mental Health Continuum Scale- Short Form (MHC-14) | Baseline
  Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
Mental Health - Mental Health Continuum Scale- Short Form (MHC-14) | 1 month - after intervention
  Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
Mental Health - Mental Health Continuum Scale- Short Form (MHC-14) | 3 month
  Mental health can be defined as a state in which an individual realizes his or her own abilities, can cope with the stresses of life, can work productively and can make a contribution,and is described by Corey L. Keyes in 3 main dimensions; emotional well being, psychological well being and social well being.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | Baseline
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. In 2006 Baer et al developed the FFMQ which consists of 39 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and non-react.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | 1 month - after intervention
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. In 2006 Baer et al developed the FFMQ which consists of 39 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and non-react.
Five Facet Mindfulness Questionnaire Short Form (FFMQ-SF) | 3 month
  Mindfulness is defined as the ability to pay attention to our own experiences without judging them. In 2006 Baer et al developed the FFMQ which consists of 39 questions that look for the 5 facets of mindfulness: observe, describe, act aware, non-judge and non-react.
Self compassion scale Short form (SCS-SF) | Baseline
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. A scale of 6 sub domains was developed and for the study, a translation of the "Self Compassion Scale Short Form - 12
Self compassion scale Short form (SCS-SF) | 1 month - after intervention
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. A scale of 6 sub domains was developed and for the study, a translation of the "Self Compassion Scale Short Form - 12
Self compassion scale Short form (SCS-SF) | 3 month
  Self compassion is understood as maintenance of full attention and opening without disconnecting from self's suffering with the desire to alleviate it in a non judgemental way, comprehending the own experience as a part of the human experience. A scale of 6 sub domains was developed and for the study, a translation of the "Self Compassion Scale Short Form - 12

CONTACTS AND LOCATIONS:
Locations (1):
- University Diego Portales, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided